CLINICAL TRIAL: NCT07153822
Title: The Multi-center, Randomized, Subject/Evaluator Blind, Active-controlled, Non-inferiority Pivotal Clinical Study to Compare the Efficacy and Safety of Collabarrier® With Guardix-sol for the Prevention of Postoperative Adhesion After Operation for Disc Herniation or Spinal Stenosis
Brief Title: Efficacy and Safety of Ionized Atelocollagen Adhesion Barrier (Collabarrier®) in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DALIM TISSEN Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRT-04
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Epidural Fibrosis; Postoperative Adhesion
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collabarrier® (Experimental)
  Interventions: Device: Collagen-based adhesion barrier
- Guardix-sol (Active Comparator)
  Interventions: Device: Sodium hyaluronate(HA) and Sodium Carboxymethylcellulose(CMC)-based adhesion barrier

INTERVENTIONS:
Device: Collagen-based adhesion barrier — Porcine Atelocollagen (Type I)
  Other Names: adhesion barrier
  Arms: Collabarrier®
Device: Sodium hyaluronate(HA) and Sodium Carboxymethylcellulose(CMC)-based adhesion barrier — Sodium Hyaluronate(HA) + Sodium Carboxymethylcellulose(CMC)
  Other Names: adhesion barrier
  Arms: Guardix-sol

SUMMARY:
This multicenter, randomized, subject- and evaluator-blinded, active-controlled, non-inferiority clinical trial was conducted to evaluate the efficacy and safety of Collabarrier®, a collagen-based adhesion barrier, compared to Guardix-sol in patients undergoing lumbar spine surgery for herniated disc or spinal stenosis.

A total of 69 adult patients scheduled for first-time partial laminectomy or discectomy were enrolled and randomly assigned to receive either Collabarrier® or Guardix-sol. The investigational device (Collabarrier®) is a gel-type atelocollagen formulation designed to prevent postoperative adhesions by acting as a physical barrier between the dura mater and surrounding tissues.

The primary outcome was the mean MRI Scar Score at 6 weeks postoperatively, assessed by independent evaluators blinded to treatment allocation. Secondary outcomes included patient-reported pain scores using a 100-mm Visual Analog Scale (VAS) for low back and leg pain, and functional limitation assessed using the Oswestry Disability Index (ODI), measured at baseline, 3 weeks, and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 19 years or older
* Patients diagnosed with lumbar disc herniation or lumbar spinal stenosis based on radiological evidence (MRI or CT) showing nerve root compression at one of the following single levels: L3-L4, L4-L5, or L5-S1
* Patients scheduled to undergo their first partial laminectomy or discectomy for the above condition
* Patients who meet at least one of the following criteria (A, B, C):
* A. Have undergone a minimum of 4 weeks of prior conservative treatment within the 6 months prior to Visit 1 (e.g., physical therapy, use of anti-inflammatory drugs, or muscle relaxants)
* B. Experience intolerable pain and are judged by the investigator to require surgery for lumbar disc herniation or spinal stenosis
* C. Have significant progression of neurological functional loss
* Patients who voluntarily provide written informed consent and are able to comply with the study procedures and visit schedule

Exclusion Criteria:

* Patients who shows alergic reaction or has previous stroke to main and other ingredients or components of the medical device for this clinical test
* Patients with a medical history of brittle bone
* Patients with a medical history of fracture in lumbar region or ligament injuries by external injury
* Patients who needs to undergo a spine surgery (osteotomy allowable) in addition to partial laminectomy or percutaneous lumbar discectomy for cure of symptom
* Patients with neurological function disorder on intestine/bladder
* Patients with any of such symptoms as excessive exudation, bleeding, acute edema and infection on the part applied
* Patients with Degenerative spinal disorder (other than disc herniation or spinal stenosis) or scoliosis (Cobb's angle is 15° or bigger)
* Patients with any of lymphatic disease, coagulation disoder and/or coagulant taken
* Patients with uncontrolled diabetes that may affect the surgery or the progress after surgery based on the tester's judgment
* Patients with desmosis or autoimmune disease or who has ever taken malignant tumor treatment within 5 years before this surgery
* Patients who has ever undergone a spine surgery on the part for this surgery
* Patients who has ever taken extradural steroid treatment within 2 weeks before surgery or oral steroid drug within 10 days before surgery
* Patients who has ever taken myelogram or lumbar puncture within 24 hours before screening
* Patients with impaired immunity or clinically significant abnormalities in clinical laboratory tests at screening Patients with immunity deteriorated or who shows clinically significant abnormality in lab test items at the moment of screening
* Patients who present clinically severe impairment in cardiovascular, digestive, respiratory, endocrine, or central nervous system, or have a mental illness that significantly affects the trial
* Participated in other clinical trials within 30 days from the screening
* A pregnant woman or lactating woman
* Patients who cannot comply with any requirement of the document form consent for this clinical test from the signing date of signature on the consent till the final day of visit
* Patients determined by the researcher to be non-conformable to this clinical trials.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Mean value of MRI scar score assessed by independent evalutor at 6 weeks after medical device use for clinical trial | 6 weeks after medical device application

SECONDARY OUTCOMES:
Mean value of 100-mm Visual Analogue Scale (VAS) for back pain assessed by the subject before and at 3 and 6 weeks after medical device use for clinical trial | Baseline, 3 weeks, and 6 weeks after medical device application
Mean value of 100-mm Visual Analogue Scale (VAS) for leg pain assessed by the subject before and at 3 and 6 weeks after medical device use for clinical trial | Baseline, 3 weeks, and 6 weeks after medical device application
Mean value of Oswestry Disability Index (ODI) for limitations of daily life assessed by the subject before and at 3 and 6 weeks after medical device use for clinical trial | Baseline, 3 weeks, and 6 weeks after medical device application

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Ajou University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor has not yet determined whether individual participant data (IPD) will be shared.